CLINICAL TRIAL: NCT01541436
Title: Remote Ischemic Preconditioning Effects on Central and Peripheral Sensitization in Healthy Volunteers-A Pilot Study
Brief Title: Remote Ischemic Preconditioning Mechanism Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 00019284
Record Dates: First submitted 2012-02-03; First posted 2012-03-01 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Remote Ischemic Preconditioning; Nociception; Central Sensitization; Peripheral Sensitization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Capsaicin, UV-B, RIPC (Active Comparator)
  Interventions: Device: Remote Ischemic Preconditioning, Capsaicin, UV-B
- Capsaicin, UV-B (Sham Comparator)
  Interventions: Device: Remote Ischemic Preconditioning, Capsaicin, UV-B

INTERVENTIONS:
Device: Remote Ischemic Preconditioning, Capsaicin, UV-B — The participants will have one disposable tourniquet applied to the left mid thigh by research personnel. The participants will then be randomized to the treatment group or sham group. The treatment group will receive 3 cycles of RIPC to the left lower leg by occluding blood flow at the thigh with a pneumatic cuff. Each cycle will consist of 5 minutes of ischemia by inflating the cuff to 300 mmHg followed by 5 minutes of reperfusion. The sham group will have the cuff inflated to no more than 15mmHg for three cycles as described above. Areas of hypersensitivity and allodynia will be obtained every 40 min for 280 min following the end of capsaicin application.

SUMMARY:
This research is being done because pain is a significant problem for patients with a variety of medical problems and following surgery or traumatic injury. Currently available pain medications may not relieve all types of pain or may relieve pain only at doses that produce side effects and potential complications.

Although Remote Ischemic Preconditioning (RIPC) appears promising, there remain several unanswered questions about how it works. This research trial will help determine how RIPC may activate the bodies natural pain control system. The goals of this study are to see if RIPC has any effect 1) on a small area of skin that will be expose to a small amount of UV- B radiation (a mild sunburn), 2) on acute thermal heat temperatures that will be applied to skin, and 3) on the sunburn-like sensation to light touch after putting capsaicin cream (the active ingredient in hot chili peppers) on skin.

Remote ischemic preconditioning is done by inflating a balloon (very similar to a blood pressure cuff) on the leg until it blocks blood flow for a few minutes. The cuff is then deflated and blood flow resumes. The process is repeated up to three times. This procedure causes the body to increase its natural pain relief system that may help to decrease the amount of postsurgical pain.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether RIPC effects peripheral sensitization, central sensitization or both and determine effect size since there is no data regarding the presumed effect. These issues cannot be easily sorted out in patients experiencing postoperative pain and hypersensitivity, since surgery affects both components. In order to address this purpose the investigators will examine, in healthy volunteers, the effect of RIPC on a manipulation which generates hypersensitivity by an exclusive peripheral mechanism (ultraviolet B (UV-B) burn) and a manipulation which generates hypersensitivity by an exclusive central mechanism (topical capsaicin). Understanding the sites at which RIPC reduces the amplification of pain after injury will be useful in determining where it would be most logically applied clinically and in guiding preclinical mechanistic studies.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers of both sexes ASA 1 or II classification
* between the ages of 18-55
* weighing less than 250 pounds
* without chronic pain
* not taking analgesics
* off caffeine for 2 days.

Exclusion Criteria:

* pregnancy
* allergy to capsaicin
* lower extremity vascular insufficiency
* active treatment for DVT
* severe thigh pain
* taking psychotropic medications, including anti-depressants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Areas of hyperalgesia and allodynia to mechanical stimuli. | 24 hours
  Hyperalgesia will be measured with vonFrey fibers and allodynia will be measured with a cotton wisp. The area will be measured in cm2.

SECONDARY OUTCOMES:
Pain intensity and unpleasantness to mechanical stimuli | 24 hours
  Using a Visual Analog Sliding Scale the intensity and unpleasantness will be measured in centimeters.
Presence of parathesias where RIPC was used | 24 hours
  After a brief tourniquet application I fully expect participants to have some degree of parasthesias. Using a standard rating scale I will record and report this.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- WakeForestUBMC, Winston-Salem, North Carolina, United States